CLINICAL TRIAL: NCT05468515
Title: Reference Interval for Pulse Oxygen Saturation in Neonates at High Altitudes During First 2 Hours and Umbilical Artery Blood Gas: a Multicenter Prospective Study
Brief Title: Reference Interval for SPO2 in Neonates at High Altitudes During First 2 Hours and Umbilical Artery Blood Gas
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-03-146-K01
Record Dates: First submitted 2022-06-13; First posted 2022-07-21 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Neonatal Disease; Altitude Hypoxia
Keywords: pulse oxygen saturation; neonate; altitude; umbilical arterial blood gas
MeSH Terms: conditions — Infant, Newborn, Diseases; Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- High altitude group: altitude level range from 2500 to 4500 meters
  Interventions: Diagnostic Test: pulse oxygen saturation
- mild altitude group: altitude level range from 500 to 2500 meters
  Interventions: Diagnostic Test: pulse oxygen saturation

INTERVENTIONS:
Diagnostic Test: pulse oxygen saturation — preductal oxygen saturation
  Other Names: umbilical blood gas analysis

SUMMARY:
Pulse oximetry offers real time and non-invasive estimation of arterial oxygen saturation in a cost-effective way, and has become a critical tool in guiding the usage of supplemental oxygen in sick newborns. During postnatal transition, pulmonary pressure decreases upon the activation of the lungs, and the ductus arteriosus constricts and closes upon the increase of partial oxygen pressure, which is negatively correlated with altitude. As a result, postnatal transition may be different at high altitudes. Umbilical cord blood gas analysis is now recommended in all high-risk deliveries because of its' value in providing information about preceding fetal hypoxic stress. But there are only limited studies about the SpO2 measurements during the first few hours after birth and umbilical blood gas analysis at high altitudes, especially at altitudes above 2500m. The primary outcome of the study is to determine the reference intervals for preductal oxygen saturation during first 2 hours of life stratified by different gestational age. The secondary outcomes is to establish the pH and lactate cutoff value of umbilical arterial blood gas at different altitude level.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a gestational age between 35 to 42 weeks who were born alive and appearing well as defined by:

  1. normal vital signs (heart rate ranging from 110 to 180 beats/minute, respiratory rate ranging from 30 to 60 breaths/minute, temperature ranging from 36.5°C to 37.5°C),
  2. absence of signs of illness such as respiratory distress.
  3. the mothers resided in the study area.

Exclusion Criteria:

* outborn, require resuscitative interventions at birth beyond blow-by oxygen,
* require admission for any reason other than observation or had a major congenital anomaly.

Ages: 0 Hours to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included infants with a gestational age between 35 to 42 weeks who were born alive and appearing well
Sampling Method: Non-Probability Sample
Enrollment: 956 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
pulse oxygen saturation | during first 2 hours after birth
  preductal pulse oxygen saturation during first two hours after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu XJ, Ma XJ, Zhao QM, Yan WL, Ge XL, Jia B, Liu F, Wu L, Ye M, Liang XC, Zhang J, Gao Y, Zhai XW, Huang GY. Pulse Oximetry and Auscultation for Congenital Heart Disease Detection. Pediatrics. 2017 Oct;140(4):e20171154. doi: 10.1542/peds.2017-1154. PMID 28939700
- [Background] Tekgunduz KS, Bilen M, Kara M, Laloglu F, Ceviz N. Oxygen saturation and perfusion index screening in neonates at high altitudes: can PDA be predicted? Eur J Pediatr. 2021 Jan;180(1):31-38. doi: 10.1007/s00431-020-03698-1. Epub 2020 Jun 5. PMID 32504134
- [Background] Gonzales GF, Salirrosas A. Arterial oxygen saturation in healthy newborns delivered at term in Cerro de Pasco (4340 m) and Lima (150 m). Reprod Biol Endocrinol. 2005 Sep 12;3:46. doi: 10.1186/1477-7827-3-46. PMID 16156890
- [Background] Zamudio S, Torricos T, Fik E, Oyala M, Echalar L, Pullockaran J, Tutino E, Martin B, Belliappa S, Balanza E, Illsley NP. Hypoglycemia and the origin of hypoxia-induced reduction in human fetal growth. PLoS One. 2010 Jan 1;5(1):e8551. doi: 10.1371/journal.pone.0008551. PMID 20049329
- [Background] Toth B, Becker A, Seelbach-Gobel B. Oxygen saturation in healthy newborn infants immediately after birth measured by pulse oximetry. Arch Gynecol Obstet. 2002 Apr;266(2):105-7. doi: 10.1007/s00404-001-0272-5. PMID 12049291
- [Background] Bakr AF, Habib HS. Normal values of pulse oximetry in newborns at high altitude. J Trop Pediatr. 2005 Jun;51(3):170-3. doi: 10.1093/tropej/fmi026. Epub 2005 Apr 26. PMID 15855304
- [Background] Ogik V, Muyingo M, Musooko M, Nankunda J. Umbilical artery lactate levels and associated maternal and newborn characteristics at Mulago National Referral Hospital: a cross-sectional observational study. BMJ Open. 2021 Aug 26;11(8):e043827. doi: 10.1136/bmjopen-2020-043827. PMID 34446476
- [Background] Bellera CA, Hanley JA. A method is presented to plan the required sample size when estimating regression-based reference limits. J Clin Epidemiol. 2007 Jun;60(6):610-5. doi: 10.1016/j.jclinepi.2006.09.004. Epub 2007 Jan 16. PMID 17493520